



# HEALTH LITERACY AND DIGITAL HEALTH IN CANCER PATIENTS «LICAPA» study

Category 3 Non-Interventional Human Research Study (RIPH 3)

## **PROTOCOL SUMMARY**

## Statistical Analysis Plan (SAP) Version n°1.0 – November 5th, 2021

Writer of the document (statisticien): Lucas Hue

Source documents: Synopsis v1.1 September 20th, 2021 Annotate CRF v1.0 September 7th, 2021

N° IB 2021-04

ID-RCB n°2021-A01725-36

This research is backed by the elderly and cancer clinical research platform (Plateforme de Recherche Clinique Personnes Agées et Cancer – PACAN)

#### **Study coordinator**

Prof. Elena PAILLAUD, PACAN Co-Coordinator,

Geriatric Department
Paris Ouest Oncogeriatrics coordination unit
Hôpital Européen Georges Pompidou
20, rue Leblanc – 75908 Paris CEDEX 15

Tél: 01.56.09.33.10 - E-mail: elena.paillaud@aphp.fr

| _ | | | | | • | | | | | | | | |
|---|----|---|---|---|---|---|---|---|---|---|---|---|----|
| • | cı | Δ | n | н | н | | m | 2 | n | 2 | Œ | Δ | rc |
| J | u | C | ш | u | ш | • | m | a | | a | s | c | ıs |

Prof. Simone MATHOULIN-PELISSIER, PACAN Coordinator,Institut BergoniéProf. Pierre-Louis SOUBEYRAN, PACAN Co-coordinator,Institut Bergonié

#### **Clinical Research and Epidemiology Unit**

Prof. Simone MATHOULIN-PELISSIER, Unit HeadInstitut BergoniéMarina PULIDO, Methodology statisticianInstitut BergoniéCaroline LALET, Clinical studies managerInstitut Bergonié

#### Inserm U1219 Epicene team

Angéline GALVIN, Epidemiologist Université Bordeaux

SPONSOR INSTITUT BERGONIÉ

229 cours de l'Argonne 33076 BORDEAUX Cedex

Tél: 05.56.33.33.33 – E-mail: drci@bordeaux.unicancer.fr

## **VERSIONS AND REVISIONS**

| Version | Date | Modification(s) | Context |
|---------|------------|-----------------|---------|
| 1.0 | 05/11/2021 | - | - |

## Table of contents

| 1. | Inti | oduc | ction | 4 |
|----|------|---------|--------------------------------------|----|
| | 1.1. | Syn | opsis (v1.1 of September 20th, 2021) | 4 |
| 2. | Obj | ectiv | res | 10 |
| | 2.1. | Prir | mary objective | 10 |
| | 2.2. | Sec | ondary objectives | 10 |
| 3. | Stu | dy or | ganisation | 10 |
| | 3.1. | Stu | dy design | 10 |
| | 3.2. | Stu | dy size | 10 |
| 4. | Def | initio | on of analysis populations | 10 |
| | 4.1. | Ana | alysis populations | 10 |
| 5. | Elig | ibility | y criteria | 11 |
| | 5.1. | Incl | lusion criteria | 11 |
| | 5.2. | Exc | lusion criteria | 11 |
| 6. | Dat | a sta | tistical analysis | 11 |
| | 6.1. | Des | scriptive methods | 11 |
| | 6.1 | 1. | Quantitative variables | 11 |
| | 6.1 | 2. | Qualitative variables | 11 |
| | 6.2. | Con | nfidence interval | 12 |
| | 6.3. | Ana | alysis methods | 12 |
| | 6.3 | 1. | Sensitivity analysis | 12 |
| | 6.3 | 2. | Exploratory analysis | 12 |
| 8. | Sta | tistica | al analysis | 12 |
| 9. | Out | com | e measures | 12 |
| | 9.1. | Prir | mary endpoint | 12 |
| | 9.2. | Sec | ondary endpoints | 13 |
| | 9.3. | Stat | tistical software | 13 |

## 1. Introduction

## 1.1. Synopsis (v1.1 of September 20th, 2021)

| TITLE | Health literacy and digital health in cancer patients |
|---|---|
| SHORT TITLE | LiCaPa |
| Sponsor | Institut Bergonié, Bordeaux |
| COORDINATOR | Prof. Elena PAILLAUD<br>Hôpital Européen Georges Pompidou, AP-HP, Paris |
| SCIENTIFIC MANAGERS | Prof. Simone MATHOULIN-PELISSIER, Institut Bergonié, Bordeaux<br>Prof. Pierre-Louis SOUBEYRAN, Institut Bergonié, Bordeaux |
| | Health literacy can be defined as « people's knowledge, motivation and competence to access, understand, appraise, and apply health information to make judgements and take decisions in everyday life concerning healthcare, disease prevention and health promotion to maintain or improve quality-of-life during the course of life ». In his literacy model, Nutbeam defines 3 skills, namely: i) functional health literacy which is sufficient basic skills in reading and writing to be able to function effectively in everyday situations, ii) communicative literacy which refers to more advanced skills which can be used to extract information and derive meaning from different forms of communication, and to apply new information to changing circumstances, and, iii) critical literacy which refers to more advanced cognitive skills which can be applied to critically analyse information, and to use this information to exert greater control over life events and situations. |
| JUSTIFICATION / BACKGROUND | In a world in which information is delivered more and more via digital tools, digital health literacy is coming to play an increasingly important part. It is based on three skills that are skills in healthcare, information skills and digital skills. Low health literacy, whether digital or not, can represent a loss of chance in terms of health [2]. Several studies have demonstrated an association between health literacy and different events such as hospitalization, understanding prescriptions, quality-of-life or even death. Given its consequences in terms of health, health literacy represents a determining element of public health, which can be acted on. In effect, taking account of health literacy is likely to improve the patient's engagement, informed decision-making and final impact on health. However, the level of health literacy is preoccupying, especially in Europe and including in France. Whereas cancers represent a high cause of morbidity and mortality worldwide, and especially in France, few studies have looked at health literacy in cancer patients and at its consequences. According to the Institut National du Cancer (Inca), cancer in the over 65s represented 62.4% of estimated cancer among all ages in 2017. |

As a result, close attention must be paid to information provided to the elderly to empower them to become fully involved in their treatment. Management of cancer in the elderly is specific due to the potential presence of various areas of fragility related to the person's age and the extent of the concomitant diseases. People age 65 and older are therefore considered among the populations likely to find themselves in difficulty due to their low level of health literacy, especially digital literacy. A pilot feasibility study was conducted in 2019 in people age 65 and over with cancer and treated in consultation or in the outpatient clinic in 6 volunteer centres in France. Overall, 72% of patients had a low level of health literacy. These results, which demonstrate low health literacy in elderly cancer patients, remain however preliminary. A larger study also including a control population of adults age 18 to 64 years is required. This multicentric transversal study will be the first to our knowledge. Health literacy in this population has never before been evaluated prospectively and the proportion presenting with a low level of health literacy was not known. **Primary objective:** Evaluate the health literacy of cancer patients using the approved French version of the Functional, Communicative and Critical Health Literary (FCCHL) scale in 2 populations: Population A: patients age 65 and over treated in an oncology or oncogeriatric outpatient clinic, or seen in an oncology or oncogeriatric consultation. Population B: young patients age 18 to 64 treated in an **OBJECTIVES** oncology or outpatient clinic, or seen in an oncology consultation. **Secondary objectives** Describe the digital health literacy of patients per population. Identify groups with low health literacy and evaluate the related factors (age, sex, lifestyle etc.) Explore the factors related to the use of the digital. Study design Multicentric, prospective, observational, transversal study Study questionnaire methodology STUDY ORGANISATION The questionnaire (Appendice 1) including: Approved French version of the FCCHL scale Questionnaire on the use of digital tools adapted from the questionnaire on digital tools, Will be completed once only. It will be completed by the participant during the oncology or oncogeriatric consultation or outpatient clinic

| | appointment, in self-questionnaire mode or face to face, assisted if necessary by a family member or member of the medical team. |
|---|---|
| | There will be no specific interview, and the patient's participation in the study shall not lead to any inconvenience or affect their treatment in any way. |
| | Expected number of centres Around 30 participating centres |
| | Around 20 participating centres. |
| | <ul> <li>Study duration</li> <li>Inclusion time: 2 weeks between September and October 2021</li> <li>Participation time for each patient: &lt; 1 hour</li> <li>Total study duration: 2 months</li> </ul> |
| RESEARCH IMPLEMENTATION | Methods of recruitment of persons questioned |
| | Patients seen in an oncology, or oncogeriatric consultation or treated in an oncology or geriatric outpatient clinic (not including full hospitalisation lasting ≥ 24h). |
| | Methods of information and tracing of consent |
| | The information leaflet (Appendice 2) will be handed to the patient by |
| | the investigator who will state the patient's consent to participate in |
| | the study in their medical record. |
| | 1. Man or woman. |
| | 2. Age ≥ 18 ans. |
| | 3. Patient treated for cancer. |
| | 4. Patient who can read and understand French. |
| INCLUSION CRITERIA | 5. Patient seen in an oncology or oncogeriatric consultation or treated |
| | in an outpatient clinic. |
| | 6. Patient in treatment or about to start treatment that has been |
| | offered to them, from the announcement consultation to 2 years after the start of treatment |
| | Patient hospitalised for longer than 24 hours. |
| EXCLUSION CRITERIA | <ol> <li>Patient nospitalised for longer than 24 hours.</li> <li>Patient with known cognitive impairment preventing them from</li> </ol> |
| | answering the questionnaire. |
| | Primary endpoint : |
| | The primary endpoint is the percentage of participants with an overall |
| | score of ≤4 on the FCCHL scale, corresponding to a low level of health |
| | literacy: |
| Outropass agraculture | <ul> <li>The FCCHL questionnaire includes 14 items, divided into 3 sub-<br/>scales, reflecting 3 health literacy skills (functional literacy,<br/>interactive literacy and critical literacy).</li> </ul> |
| OUTCOMES MEASURES | The FCCHL is validated and a French translation is available |
| | The scores for the tree sub-scales are described for each |
| | population, and an overall score will be calculated by |
| | determining the mean score of the 3 sub-scales. |
| | <ul> <li>An overall score of ≤4 points to a low level of literacy.</li> </ul> |
| | · |
| | Secondary endpoints: The secondary endpoints include: |

- The questionnaire on the use of digital tools will be described per item :
  - o This questionnaire includes 10 items.
  - A Likert-type scale with five modalities of response is proposed (never, rarely, sometimes, often, always).
  - No overall score will be calculated.
  - The responses to the FCCHL scales and to the questionnaire on the use of digital will also be described by sub-groups defined according to the patient's characteristics at baseline (age, sex, lifestyle, etc.)

#### Total: 840 patients

Population A: 420 patientsPopulation B: 420 patients

## The primary endpoint is the percentage of participants with an overall score of ≤4 on the FCCHL scale, evaluated in 2 populations:

- Population A: patients age 65 and over treated in an oncology or oncogeriatric outpatient clinic, or seen in an oncology or oncogeriatric consultation.
- Population B: young patients age 18 to 64 treated in an oncology or outpatient clinic or seen in an oncology consultation.

We plan to include around 300 eligible and assessable patients (overall score available) for the primary endpoint in each of the two populations (A and B). A total of 420 patients per populations will be included in this study in order to take account of 40% of non-eligible/non-assessable patients (score not available - 35% of patients had not fully completed the questionnaire in the feasibility study).

Inclusions will last 2 whole weeks, between September and October 2021, in 21 centres which will include at least 40 patients each.

Our primary objective is to describe the percentage of patients with low health literacy, corresponding to an overall score of ≤4 on the FCCHL scale. We found an overall score of ≤4 for 72% of the patients in our feasibility study. Also, according to the latest report from the OECD, 60% of French adults have a low level of literacy. Finally, around 88% of the elderly in Canada have a low level of health literacy compared to 60% of adults.

In each of the two populations, presuming 300 subjects are recruited for whom the overall score will be available, below we provide the precision of the estimations according to the expected percentage of subjects with a low level of literacy, between 60% and 90%. This percentage was calculated using the Wald test (normal approximation) (NQuery).

#### **S**TUDY SIZE

| | Expected | | | 95% confidence interval |
|---|---|---|---|---|
| | percenta | Precision | CI width | (95%CI) |
| | ge | | | (557661) |
| | 60% | 5.5% | 11% | [54.5% ; 65.5%] |
| | 70% | 5.2% | 10.4% | [64.8% ; 75.2%] |
| | 80% | 4.5% | 9% | [75.5% ; 84.5%] |
| | 90% | 3.4% | 6.8% | [86.6 % ; 93.4%] |
| | Analysis popu | lations: | | |
| | deviation of Eligible a completed health lite Primary endpo The primary population The analyst population The perce be calculated be calculated be a population. | from the eligand assessand all 14 items racy score. Soint analysis ary endpoint analysis ary endpoint analysis ary endpoint and B. The ses will be cons A and B. The ses are as follow tem on the Fach patient, | sibility crite<br>ble popula<br>s on the FC<br>:<br>analysis w<br>onducted in<br>tients with<br>as:<br>CCHL takes<br>a literacy | etion: eligible patients having CHL scale to calculate the overall vill cover the eligible, assessable independently in each of the two a low level of health literacy will a score of 1 to 5 points. score per sub-scale (functional, |
| DATA STATISTICAL ANALYSIS | number scale. An over determined literace of the performance of elignature and the sinteractive of the quantistandard of the responsible of the quantistandard of the quality of the qual | er of points The score ca erall literacy mining the m y scores. The ercentage of e calculated er of patient gible and as ed along wit onses to the n (A, B) by su tandard-dev e, critical and itative variab deviation if other deso ative variable | divided by an range fro score will be easore can a patients who for each pus with an obsessable push its 95% coe FCCHL so be scale and iation of the assumation of the assumat | the determined by calculating the the number of items on the subsem 1 to 5. The calculated for each patient, by functional, interactive and critical range from 1 to 5. With a low level of health literacy opulation (A, B), by dividing the verall score of ≤4 by the number atients. The percentage will be confidence interval (binomial law). Cale will be described for each diversall, by calculating the mean the 4 literacy scores (functional, sulting for each patient. Described based on the mean and aption of normality is followed, tistics will be used (minimum, described based on numbers and a percentage (%). |
| EXPECTED RESULTS | For patients:<br>Determining t | he level of | health lite | eracy of cancer patients, with a d make it possible to provide |

information that is more compatible with the mean level of literacy in this population. Determining the level of digital health literacy in the same population would make it possible to find out whether digital follow-up is feasible. Appropriate education could be implemented to develop their ability to access, understand, appraise, and apply basic health information.

#### For public health:

Better understanding of health literacy would make it possible to improve and develop prevention actions for cancer patients and elderly patients in particular. This could lead to a decrease in healthcare costs, better treatment compliance, reduction in adverse effects and fewer hospitalisations, emergency department admissions and readmissions.

#### 2. Objectives

#### 2.1. Primary objective

Evaluate the health literacy of cancer patients using the approved French version of the Functional, Communicative and Critical Health Literacy (FCCHL) scale in 2 populations:

- Population A: patients age 65 and over treated in an oncology or oncogeriatric outpatient clinic, or seen in an oncology or oncogeriatric consultation.
- Population B: young patients age 18 to 64 treated in an oncology or outpatient clinic, or seen in an oncology consultation.

#### 2.2. Secondary objectives

- Describe the digital health literacy of patients per population.
- Identify groups with low health literacy and evaluate the related factors (age, sex, lifestyle etc.).
- Explore the factors related to the use of the digital.

#### 3. Study organisation

#### 3.1. Study design

• Multicentric, prospective, observational, transversal study.

#### 3.2. Study size

• Total: 840 patients

Population A: 420 patientsPopulation B: 420 patients

The primary endpoint is the percentage of participants with an overall score of ≤4 on the FCCHL scale, evaluated in 2 populations.

- Population A: patients age 65 and over treated in an oncology or oncogeriatric outpatient clinic, or seen in an oncology or oncogeriatric consultation.
- Population B: young patients age 18 to 64 treated in an oncology or outpatient clinic, or seen in an oncology consultation.
- We plan to include around 300 eligible and assessable patients (overall score available) for the primary endpoint in each of the two populations (A and B). A total of 420 patients per population will be included in this study in order to take account of 40% of non-eligible/non-assessable patients (score not available 35%) of patients had not fully completed the questionnaire in the feasibility study).

### 4. Definition of analysis populations

#### 4.1. Analysis populations

Eligible population: all the patients included without major deviation from the eligibility criteria.

**Eligible and assessable population**: eligible patients having a completed all 14 items on the FCCHL scale to calculate the overall health literacy score.

## 5. Eligibility criteria

#### 5.1. Inclusion criteria

| Criteria | eFORM<br>variable | Control |
|---|---|---|
| 1. Man or women | SEXE | <b>SEXE</b> in (1 2) |
| 2. Age ≥ 18 years | AGE | AGE ge 18 |
| 3. Patient treated for cancer | LOC_CANX | X= 1 à 21<br>LOC_CANX=1 or<br>LOC_CANX=1 |
| 4. Patient who can read and understand French | NA | Investigator decision |
| 5. Patient seen in an oncology or oncogeriatric consultation or treated in an outpatient clinic. | LIEU | <b>LIEU</b> in (1 2 3) |
| 6. Patient in treatment or about to start treatment that has been offered to tem, from the announcement consultation to 2 years after the start of treatment | TRT_CAN1 TRT_CAN2 TRT_CAN3 TRT_CAN4 TRT_CAN5 TRT_CAN6 TRT_CAN7 TRT_CAN8 | TRT_CAN1=1 or TRT_CAN2=1 or TRT_CAN3=1 or TRT_CAN4=1 or TRT_CAN5=1 or TRT_CAN6=1 or TRT_CAN7=1 or TRT_CAN8=1 |

#### 5.2. Exclusion criteria

| Criteria | eFORM<br>variable | Control |
|---|---|---|
| 1. Patient hospitalised for longer than 24 hours. | NA | Investigator decision |
| <ol><li>Patient with known cognitive<br/>impairment preventing them<br/>from answering the questionnaire</li></ol> | NA | Investigator decision |

<sup>\*</sup>NA: not applicable

## 6. Data statistical analysis

#### 6.1. Descriptive methods

#### 6.1.1. Quantitative variables

Quantitative variables will be described based on the mean and standard-deviation if the assumption of normality is followed, otherwise other descriptive statistics will be used (minimum, maximum, median and quartile)

#### 6.1.2. Qualitative variables

The qualitative variables will be described base on numbers and associated frequencies, given as a percentage (%).

#### 6.2. Confidence interval

The percentage of patients with a low level of health literacy will be reported along with its 95% confidence interval (binomial lax).

#### 6.3. Analysis methods

#### 6.3.1. Sensitivity analysis

Sensitivity analyses could be carried out by varying the discrimination threshold for a low level of health literacy (currently global score  $\leq 4 =$  low level of literacy).

#### 6.3.2. Exploratory analysis

Statistical tests will be carried out (chi-square test or Fisher's exact test) to analyse the associations between low health literacy and patient characteristics at inclusion. Univariate and multivariate analyses will also be carried out.

#### 8. Statistical analysis

#### **Analysis population:**

- Eligible population: all the patients included without major deviation from the eligibility criteria.
- Eligible and assessable population: eligible patients having completed all 14 items on the FCCHL scale to calculate the overall health literacy score.

#### Primary endpoint analysis:

- The primary endpoint analysis will cover the eligible, assessable population.
- The analyses will be conducted independently in each of the two populations A and B.
- The percentage of patients with a low level of health literacy will be calculated as follows:
  - o Each item on the FCCHL takes a score of 1 to 5 points.
  - For each patient, a literacy score per sub-scale (functional, interactive and critical) will be determined by calculating the number of points divided by the number of items on the subscale. The score can range from 1 to 5.
  - An overall literacy score will be calculated for each patient, by determining the mean of the functional, interactive and critical literacy scores. The score can range from 1 to 5.
  - o The percentage of patients with a low level of health literacy will be calculated for each population (A, B), by diving the number of patients with an overall score of ≤4 by the number of eligible and assessable patients. The percentage will be reported along with its 95% confidence interval (binomial law).
- The responses to the FCCHL scale will be described for each population (A, B) by sub-scale and overall, by calculating the mean and the standard-deviation of the 4 literacy scores (functional; interactive, critical and overall) resulting for each patient.
- The quantitative variables will be described based on the mean and standard-deviation if the assumption of normality is followed, otherwise other descriptive statistics will be used (minimum, maximum, median and quartile).
- The qualitative variables will be described based on numbers and associated frequencies, given as a percentage (%).

#### 9. Outcome measures

#### 9.1. Primary endpoint

The primary endpoint is the percentage of participants with an overall score of ≤4 on the FCCHL scale, corresponding to a low level of health literacy:

- The FCCHL questionnaire includes 14 items, divided into 3 sub-scales, reflection 3 health literacy skills (functional literacy, interactive literacy and critical literacy).
- The FCCHL is validated and a French translation is available.
- The score for the tree sub-scales are described for each population, and an overall score will be calculated by determining the mean score for the 3 sub-scales.
- An overall score of ≤4 points to a low level of literacy

| Criteria | eFORM<br>variable | SAS code |
|---|---|---|
| Percentage of patients with an overall score ≤4 on the FCCHL scale corresponding to a low level of health literacy | | <pre>SCORE_GLO = mean(score_fonc, score_int, score cri) TAUX=SCORE_GLO/EVA</pre> |

#### 9.2. Secondary endpoints

The secondary endpoints include:

- The questionnaire on the use of digital tools will be described per item:
  - o This questionnaire includes 10 items.
  - A Likert-type scale with five modalities of response is proposed (never, rarely, sometimes, often, always).
  - No overall score will be calculated
- The responses to the FCCHL scales and to the questionnaire on the use of the digital will also be described by sub-groups defined according to the patient's characteristics at baseline (age, sex, lifestyle, etc.).

#### 9.3. Statistical software

The main statistical analyses will be performed using SAS v9.4. Other statistical software to produce graphics, for example, could be used.

## Appendice 1

#### **CREATION OF A NEW INDICATOR VARIABLE**

Patients fulfilling inclusions and non-inclusion criteria will be considered as ELIGIBLE (ELI = 1).

**New binary variable ELI** 

Label: "Eligible population"

ELI = 1 if the patient is eligible

ELI = 0 if the patient is not eligible

| Criteria | eFORM<br>variable | Control |
|---|---|---|
| Eligible population | C1I C2I C3I C4I C5I C6I C1NI<br>C2NI | C1I NE 0 and C2I NE 0 and C3I<br>NE 0 and C4I NE 0 and C5I NE 0<br>and C6I NE 0<br>AND<br>C1NI NE 1 and C2NI NE 1 |

## Appendice 2

#### **CREATION OF A NEW INDICATOR VARIABLE**

Patients fulfilling all 14 items of FCCHL scale will be considered as ASSESSABLE (EVA=1).

#### **Variable binaire EVA**

Label: "Assessable Population"

EVA= 1 if the patient is included in assessable population
EVA= 0 if the patient is not included in assessable population

| Criteria | eFORM<br>variable | Control |
|---|---|---|
| Eligible population | ELI | ELI = 1<br>AND |
| Assessable population | EVA NOT_MOT NOT_ECR NOT_CONT NOT_TPS NOT_LIRE INF_SOU INF_DIS INF_OBT INF_MED INF_QUO TRT_INF TRT_CRE TRT_COR TRT DEC | NOT_MOT ne . and NOT_ECR ne . and NOT_CONT ne . and NOT_TPS ne . and NOT_LIRE ne . and INF_SOU ne . and INF_DIS ne . and INF_OBT ne . and INF_MED ne . and INF_QUO ne . and TRT_INF ne . and TRT_CRE ne . and TRT_COR ne . and TRT_DEC ne . Then EVA=1 Else EVA=0 |